CLINICAL TRIAL: NCT06929065
Title: Randomized Prospective Trial of Focal Therapy (HIFU vs Cryo) for Early Stage Unifocal Prostate Cancer
Brief Title: Randomized Trial of HIFU vs. Cryo for Prostate Cancer
Acronym: KPFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Principal Investigator, David S Finley, MD, PI, Kaiser Permanente
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KPFT
Record Dates: First submitted 2022-11-16; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer; Prostate Cancer Stage I; Prostate Cancer Stage II; High Intensity Focused Ultrasound; HIFU; Cryoablation
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized prospective open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HIFU (Experimental): HIFU
  Interventions: Procedure: HIFU vs Cryoablation
- Cryoablation (Active Comparator): Cryo
  Interventions: Procedure: HIFU vs Cryoablation

INTERVENTIONS:
Procedure: HIFU vs Cryoablation — HIFU vs cryoablation

SUMMARY:
HIFU has been FDA approved and is widely utilized across the United States and Europe for the treatment of prostate cancer. Despite this, HIFU has not been offered within SCPMG until now due to growing patient demand. We have offered cryoablation. This pilot study will determine the efficacy of HIFU vs. cryoablation focal therapy for early stage prostate cancer within SCPMG. We hope to elucidate whether outcomes are similar between the two modalities.

DETAILED DESCRIPTION:
All men presenting with elevated prostate specific antigen (PSA) will be required to undergo an initial multiparametric MRI (MRI) and 14 core systematic biopsy. Decipher genomic testing will be run on all prostate cancer specimens. 48 men with with unifocal low-intermediate risk prostate cancer (clinical stage T1-T2, Gleason group 1-2) prostate cancer will be offered focal therapy vs. conventional therapy (surgery or radiation) via shared decision making. Those who elect focal therapy (FT) will be enrolled and randomized 1:1 to HIFU or cryoablation. Men with negative biopsy, multifocal disease, or unfavorable intermediate risk or higher disease will be excluded and offered standard therapy (surgery or radiation).

Following treatment, mpMRI and biopsy will be performed at 3mo. Baseline, 3mo, 6mo and 12mo post-treatment PSA will be obtained. In field and out of field cancer recurrence will be determined. Baseline and 3mo American Urologic Association Symptom Score (AUAss) and International Index of Erectile Function (IIEF) will be recorded as well as any treatment related side-effects or complications. SpaceOAR hydrogel will be utilized for all posterior lesions.

ELIGIBILITY:
Inclusion Criteria:

1. All men age 40 or older with Gleason group 1 or 2 prostate cancer involving a single or adjacent sextants
2. PSA < 10
3. mpMRI without extracapsular extension or seminal vesicle invasion (non-focal MRI or organ confined)
4. mpMRI which is either nonfocal or concordant with biopsy.

Exclusion Criteria:

1. Gleason group 3 or higher
2. Multifocal disease
3. mpMRI with ECE or SVI
4. PSA > 10
5. Active anorectal disease
6. Age > 80

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
In-field cancer persistence | 3 months
  MRI and biopsy results

SECONDARY OUTCOMES:
AUAss change from baseline | month 3, month 6, month 12, month 24
  Change in urination over
IIEF change from baseline | month 3, month 6, month 12, month 24
  Change in sexual function over time
Complications and satisfaction | month 3, month 6, month 12, month 24
PSA | month 3, month 6, month 12, month 24
  PSA change over time

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bakavicius A, Marra G, Macek P, Robertson C, Abreu AL, George AK, Malavaud B, Coloby P, Rischmann P, Moschini M, Rastinehad AR, Sidana A, Stabile A, Tourinho-Barbosa R, de la Rosette J, Ahmed H, Polascik T, Cathelineau X, Sanchez-Salas R. Available evidence on HIFU for focal treatment of prostate cancer: a systematic review. Int Braz J Urol. 2022 Mar-Apr;48(2):263-274. doi: 10.1590/S1677-5538.IBJU.2021.0091. PMID 34003610
- [Background] Guillaumier S, Peters M, Arya M, Afzal N, Charman S, Dudderidge T, Hosking-Jervis F, Hindley RG, Lewi H, McCartan N, Moore CM, Nigam R, Ogden C, Persad R, Shah K, van der Meulen J, Virdi J, Winkler M, Emberton M, Ahmed HU. A Multicentre Study of 5-year Outcomes Following Focal Therapy in Treating Clinically Significant Nonmetastatic Prostate Cancer. Eur Urol. 2018 Oct;74(4):422-429. doi: 10.1016/j.eururo.2018.06.006. Epub 2018 Jun 28. PMID 29960750
- [Background] von Hardenberg J, Westhoff N, Baumunk D, Hausmann D, Martini T, Marx A, Porubsky S, Schostak M, Michel MS, Ritter M. Prostate cancer treatment by the latest focal HIFU device with MRI/TRUS-fusion control biopsies: A prospective evaluation. Urol Oncol. 2018 Sep;36(9):401.e1-401.e9. doi: 10.1016/j.urolonc.2018.05.022. Epub 2018 Aug 6. PMID 30093211
- [Background] Westhoff N, Ernst R, Kowalewski KF, Schmidt L, Worst TS, Michel MS, von Hardenberg J. Treatment decision satisfaction and regret after focal HIFU for localized prostate cancer. World J Urol. 2021 Apr;39(4):1121-1129. doi: 10.1007/s00345-020-03301-0. Epub 2020 Jun 12. PMID 32533247
- [Background] Lovegrove CE, Peters M, Guillaumier S, Arya M, Afzal N, Dudderidge T, Hosking-Jervis F, Hindley RG, Lewi H, McCartan N, Moore CM, Nigam R, Ogden C, Persad R, Virdi J, Winkler M, Emberton M, Ahmed HU, Shah TT, Minhas S. Evaluation of functional outcomes after a second focal high-intensity focused ultrasonography (HIFU) procedure in men with primary localized, non-metastatic prostate cancer: results from the HIFU Evaluation and Assessment of Treatment (HEAT) registry. BJU Int. 2020 Jun;125(6):853-860. doi: 10.1111/bju.15004. Epub 2020 Feb 11. PMID 31971335
- [Background] Connor MJ, Gorin MA, Ahmed HU, Nigam R. Focal therapy for localized prostate cancer in the era of routine multi-parametric MRI. Prostate Cancer Prostatic Dis. 2020 Jun;23(2):232-243. doi: 10.1038/s41391-020-0206-6. Epub 2020 Feb 12. PMID 32051551
- [Background] Biermann K, Montironi R, Lopez-Beltran A, Zhang S, Cheng L. Histopathological findings after treatment of prostate cancer using high-intensity focused ultrasound (HIFU). Prostate. 2010 Aug;70(11):1196-200. doi: 10.1002/pros.21154. PMID 20564422
- [Background] van Velthoven R, Aoun F, Marcelis Q, Albisinni S, Zanaty M, Lemort M, Peltier A, Limani K. A prospective clinical trial of HIFU hemiablation for clinically localized prostate cancer. Prostate Cancer Prostatic Dis. 2016 Mar;19(1):79-83. doi: 10.1038/pcan.2015.55. Epub 2015 Nov 24. PMID 26597660
- [Background] Hamdy FC, Elliott D, le Conte S, Davies LC, Burns RM, Thomson C, Gray R, Wolstenholme J, Donovan JL, Fitzpatrick R, Verrill C, Gleeson F, Singh S, Rosario D, Catto JW, Brewster S, Dudderidge T, Hindley R, Emara A, Sooriakumaran P, Ahmed HU, Leslie TA. Partial ablation versus radical prostatectomy in intermediate-risk prostate cancer: the PART feasibility RCT. Health Technol Assess. 2018 Sep;22(52):1-96. doi: 10.3310/hta22520. PMID 30264692
- [Background] Chin JL, Al-Zahrani AA, Autran-Gomez AM, Williams AK, Bauman G. Extended followup oncologic outcome of randomized trial between cryoablation and external beam therapy for locally advanced prostate cancer (T2c-T3b). J Urol. 2012 Oct;188(4):1170-5. doi: 10.1016/j.juro.2012.06.014. Epub 2012 Aug 15. PMID 22901586
- [Background] Donnelly BJ, Saliken JC, Brasher PM, Ernst SD, Rewcastle JC, Lau H, Robinson J, Trpkov K. A randomized trial of external beam radiotherapy versus cryoablation in patients with localized prostate cancer. Cancer. 2010 Jan 15;116(2):323-30. doi: 10.1002/cncr.24779. PMID 19937954